CLINICAL TRIAL: NCT03298009
Title: Subclinical Inflammation, Myocardial Function and Fatty Acid Metabolism in Patients With Type 2 Diabetes and Heart Failure: Impact of a Short-term Treatment With Canagliflozin - a Pilot Study
Brief Title: Impact of a Short-term Treatment With Canagliflozin (Canacardia-HF)
Acronym: Canacardia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: end of contract negociations
Sponsor: Université de Sherbrooke (Other)
Collaborators: Janssen Inc. (Industry)
Responsible Party: Principal Investigator, André Carpentier, tenured professor, Université de Sherbrooke
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 28431754DIA4029
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Type2 Diabetes; Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Canagliflozin; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, double-blind, randomized crossover 2-week intervention study.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment 1 (Placebo Comparator): placebo oral capsule will be administered once daily, for 2 weeks
  Interventions: Drug: Placebo oral capsule; Radiation: PET imaging
- Treatment 2 (Experimental): Canagliflozine 100mg once daily, for 2 weeks
  Interventions: Drug: Canagliflozin 100mg; Radiation: PET imaging

INTERVENTIONS:
Drug: Canagliflozin 100mg — 2-week intervention
  Other Names: Invokana
  Arms: Treatment 2
Drug: Placebo oral capsule — 2-week intervention
  Arms: Treatment 1
Radiation: PET imaging — 1 day postprandial metabolic protocol at the end of treatment: CT scan followed by dynamic and pancorporel imaging

SUMMARY:
It is a mechanistic proof-of-concept study to demonstrate how SGLT-2 inhibitors (Canagliflozin) may have a beneficial role on cardiac energetic efficiency.

Patients with type 2 diabetes and with HF diagnosed for at least 3 months will be selected. The participants will be randomized to a double-blind, crossover 2-week placebo vs. Cana 100 mg once daily, an interventional trial with a one-month washout period in between.

At the term of the two-week placebo and canagliflozin treatment periods (visits 2 and 4), each participant will undergo an identical postprandial metabolic study with positron emission tomography (PET) and stable isotopic tracer methods.

DETAILED DESCRIPTION:
Non-invasive Positron Emission Tomography (PET) imaging method allows to measure myocardial uptake and organ-specific partitioning of dietary fatty acids (DFA). It allows to study kidney, liver, skeletal muscles and adipose tissues DFA utilization, whole body fatty acid turnover and oxidation rates, myocardial oxidative metabolism and left ventricular (LV) function that are other likely targets of SGLT-2 inhibitors. Thus, the PET is ideal to verify the very interesting hypothesis that, increase in liver fatty acid utilization and/or adipose tissue dietary fatty acid uptake, may lead to reduced cardiac utilization of fatty acids and improved cardiac energetic efficiency.

.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c 7.5 -10.5%;
* LVEF < 40%;
* NYHA class 2 or 3;
* NT pro-BNP level > 600 pg/mL;
* Being on a stable-dose metformin therapy max 2500 mg/day or other hypoglycemic therapy and RAAS-blocking agents for at least 8 weeks;
* Being on optimal and stable-doses of heart failure medication including diuretics for at least 4 weeks;

Exclusion Criteria:

* age <18 yo;
* NYHA class 4;
* Treatment with a fibrate or thiazolidinedione;
* Unstable or advanced renal failure;
* Unstable or new medical or surgical condition within the past 3 months;
* Heart failure caused by active inflammatory condition such as sarcoidosis or any form of myocarditis;
* History of diabetic ketoacidosis;
* Not on a stable regimen for at least 8 weeks before the screening visit;
* Female of child-bearing potential who is pregnant, breast feeding or intends to become pregnant or pre-menopausal female with a positive serum pregnancy test at the time of enrollment;
* Patients post bariatric surgery, or on weight loss medication;
* Contraindications to metformin, including allergy or intolerance;
* Hospitalization for heart failure within the 60 days prior to enrollment;
* Admission for an acute coronary syndrome, percutaneous coronary intervention, or cardiac surgery within the 60 days prior to enrollment;
* Planned cardiovascular revascularization (percutaneous intervention or surgical) or major cardiac surgery (coronary artery bypass grafting, valve replacement, ventricular assist device, cardiac transplantation, or any other surgery requiring thoracotomy) within the 90 days after enrollment;
* Patients who are volume depleted based upon physical examination at the time of enrollment;
* Chronic disabling illness;
* History of substance abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Change to be observed with canagliflozin on myocardial dietary fatty acid uptake | 3 months
  will be assessed using oral administration of 18-fluoro-thiaheptadecanoic acid ([18F]-FTHA) with sequential dynamic.
  PET/CT scanning.
Change to be observed with canagliflozin on whole-body partitioning. | 3 months
  will be assessed using oral administration of 18-fluoro-thiaheptadecanoic acid ([18F]-FTHA, with static PET/CT scanning

SECONDARY OUTCOMES:
myocardial and liver NEFA uptake | 3 months
  using PET with [11C]-palmitate
NEFA oxidative rate | 3 months
  using PET with [11C]-acetate
plasma NEFA turnover | 1 year
  using i.v. infusion of [U-13C]-palmitate

OTHER OUTCOMES:
Insulin sensitivity | 1 year
  will be determined using the HOMA-IR (based on fasting insulin and glucose levels)
Insulin secretion rate | 1 year
  will be assessed using deconvolution of plasma C-peptide with standard Cpeptide kinetic parameters
β-cell function | 1 year
  will be assessed by calculation of the disposition index (DI) that is insulin secretion in response to the ambient insulin
hormonal response | 1 year
  will be determined using a multiplex assay system
Biomarkers | 1 year
  Assays will be performed using the BIOPLEX
body composition | 3 months
  DXA

CONTACTS AND LOCATIONS:
Overall Officials: André C. Carpentier, Principal Investigator — Université de Sherbrooke